CLINICAL TRIAL: NCT01061099
Title: A Pilot Study to Assess the Safety and Feasibility of Repeated Infusions of Mesenchymal Stromal Cells (MSC) in Children With Osteogenesis Imperfecta
Brief Title: Repeated Infusions of Mesenchymal Stromal Cells in Children With Osteogenesis Imperfecta
Acronym: STOD3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Edwin Horwitz, Attending Physician, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-4-5947
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Osteogenesis Imperfecta Type II; Osteogenesis Imperfecta Type III
Keywords: Type II or Type III Osteogenesis imperfecta; OI; Mesenchymal Stromal Cells; MSC
MeSH Terms: conditions — Osteogenesis Imperfecta; Osteogenesis imperfecta, type 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stratum A (Active Comparator): Subjects with a diagnosis of Type II or Type III osteogenesis imperfecta who have previously undergone a bone marrow transplant. Intervention: Mesenchymal Stromal Cells.
  Interventions: Biological: Mesenchymal Stromal Cells
- Stratum B (Active Comparator): Subjects with Type II or III osteogenesis imperfecta who have not undergone a bone marrow transplant. Intervention: Mesenchymal Stromal Cells.
  Interventions: Biological: Mesenchymal Stromal Cells

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells — Both cohorts will receive multiple infusions of ex-vivo expanded MSCs. Stratum A may use previously harvested and cryopreserved bone marrow mononuclear cells from original BMT donor or freshly harvested or cryopreserved bone marrow mononuclear cells obtained from a haploidentical healthy parent or sibling. Stratum B will only receive freshly harvested or cryopreserved bone marrow
  Other Names: ex-vivo expanded MSCs

SUMMARY:
This is a study to evaluate the safety and effectiveness of repeated Mesenchymal Stromal Cells (MSC) infusions to patients with Type II or III osteogenesis imperfecta (OI).

Participants will receive MSC infusions approximately every 4 months to complete a total of 6 infusions over 20 months. Participants will be followed for 4 months post their last MSC infusion.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the safety and efficacy of repeated MSC infusions to subjects with OI. This study will evaluate subjects on two separate strata. Stratum A will include subjects with a diagnosis of Type II or Type III osteogenesis imperfecta who have previously undergone a bone marrow transplant. Stratum A may use previously harvested and cryopreserved bone marrow mononuclear cells from original BMT donor or freshly harvested or cryopreserved bone marrow mononuclear cells obtained from a haploidentical healthy parent or sibling. Stratum B will include subjects with Type II or III osteogenesis imperfecta who have not undergone a bone marrow transplant. Stratum B will only receive freshly harvested or cryopreserved bone marrow mononuclear cells from a haploidentical healthy parent or sibling.

Participants will receive MSC infusions approximately every 4 months to complete a total of 6 infusions over 20 months. Participants will be followed for 12 months post their last MSC infusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects less than or equal to 19 years of age at the time of enrollment
* Children with a diagnosis of severe of Type II or III osteogenesis imperfecta
* Parent or sibling greater than or equal to 18 years of age, donor willing to or has already undergone HLA typing, and willing and able to provide bone marrow
* BMT greater than 5 years ago for Stratum A

Exclusion Criteria:

* Dependent on supplemental oxygen
* Concurrent Infection

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To determine the safety or repeated infusions of donor-derived and MSCs in subjects with severe osteogenesis imperfecta > 5years after an allogeneic bone marrow transplant and no prior bone marrow transplant. | Completion of study

SECONDARY OUTCOMES:
To determine if MSCs elicit an immune response after repeated infusions. | Completion of study
To determine the change in clinical course (growth, bone mineral content, fracture rate, development/activities) of subjects after experimental MSC intervention therapy as compared with each subject's own pre-MSC intervention therapy. | Completion of Study

CONTACTS AND LOCATIONS:
Overall Officials: Alix Seif, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Horwitz EM, Gordon PL, Koo WK, Marx JC, Neel MD, McNall RY, Muul L, Hofmann T. Isolated allogeneic bone marrow-derived mesenchymal cells engraft and stimulate growth in children with osteogenesis imperfecta: Implications for cell therapy of bone. Proc Natl Acad Sci U S A. 2002 Jun 25;99(13):8932-7. doi: 10.1073/pnas.132252399. PMID 12084934
- [Background] Horwitz EM, Prockop DJ, Gordon PL, Koo WW, Fitzpatrick LA, Neel MD, McCarville ME, Orchard PJ, Pyeritz RE, Brenner MK. Clinical responses to bone marrow transplantation in children with severe osteogenesis imperfecta. Blood. 2001 Mar 1;97(5):1227-31. doi: 10.1182/blood.v97.5.1227. PMID 11222364
- [Background] Horwitz EM, Prockop DJ, Fitzpatrick LA, Koo WW, Gordon PL, Neel M, Sussman M, Orchard P, Marx JC, Pyeritz RE, Brenner MK. Transplantability and therapeutic effects of bone marrow-derived mesenchymal cells in children with osteogenesis imperfecta. Nat Med. 1999 Mar;5(3):309-13. doi: 10.1038/6529. PMID 10086387